CLINICAL TRIAL: NCT00804518
Title: Aerobic Interval Training Reduces and Compensates Age Related Decline in Cardiac Function
Brief Title: Effect of Exercise on Heart Function in Healthy Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4.2008.2177
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Diastolic Dysfunction
Keywords: Aging; Diastolic dysfunction; Systolic function; Exercise; Echocardiography; tissue Doppler imaging; Cardiac function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise intervention (Experimental)
  Interventions: Other: Aerobic interval training

INTERVENTIONS:
Other: Aerobic interval training — High intensity aerobic interval training consists of 10 minutes warm up at ~60% of maximal heart rate, 4x4 minutes intervals at 90-95 % of maximal heart rate corresponding to 85-90% of VO2max) walking/running uphill on a treadmill, with three minutes active pause between the exercise bouts at 60-70% maximal heart rate. The session is terminated with 3 minutes cool down. Total exercise time is 38 minutes.The training is supervised by an exercise physiologist and the subjects train 3 times per week for 12 weeks.

SUMMARY:
The purpose of this study is to determine the effect of aerobic interval training on left- and right ventricular diastolic- and systolic function on healthy, sedate people over 70 years. The old sedate cohort will be compared to young, sedate subjects also performing aerobic interval training and old master athletes without intervention.

DETAILED DESCRIPTION:
Aging is associated with a reduced diastolic and systolic function of the heart. Earlier studies have shown that physical exercise can improve both systolic and diastolic function. However the impact on age-related cardiac function is to some extent conflicting. The use of different training intensities will impact on the cardiac result. We have in earlier studies shown aerobic interval training at 90 % of maximal heart rate (4x4 minutes) to have more impact on cardiac function, endothelial function and maximal oxygen uptake compared to moderate intensity.

To our knowledge the effect of aerobic interval training on cardiac function has not been studied in an old, sedate group before.

ELIGIBILITY:
Inclusion Criteria:

* over 70 years, healthy
* not exercising more than twice per week

Exclusion Criteria:

* chronic illness
* chronic use of any medication
* regular smoking
* metabolic or cardiovascular diseases

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Improvement of left and right ventricular early diastolic tissue velocity at rest and sub maximal exercise ,e'. | 12 weeks

SECONDARY OUTCOMES:
Improvement of left and right ventricular systolic tissue velocity function at rest and sub maximal exercise, S'. | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bjork Ingul, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- Ntnu/Dmf/Isb, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Molmen HE, Wisloff U, Aamot IL, Stoylen A, Ingul CB. Aerobic interval training compensates age related decline in cardiac function. Scand Cardiovasc J. 2012 Jun;46(3):163-71. doi: 10.3109/14017431.2012.660192. Epub 2012 Feb 20. PMID 22273242